CLINICAL TRIAL: NCT06679335
Title: Examining the Effect of Lateralization Imagery Training on EEG Brain Oscillations, Pain Intensity, Proprioception, Kinesiophobia and Body Awareness in Individuals With Chronic Neck Pain
Brief Title: Examining the Effect of Lateralization Imagery Training on EEG Brain Oscillations in Individuals With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Aysegul Bostan, Lecturer, Bahçeşehir University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAU-AYSEGULBOSTAN-001
Record Dates: First submitted 2024-06-12; First posted 2024-11-07 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Neck Pain
Keywords: Chronic Neck Pain; Lateralization Imagery Training; EEG Brain Oscillations; Proprioception; Body Awareness
MeSH Terms: conditions — Chronic Pain; Neck Pain

STUDY DESIGN:
Intervention Model Description: Both healthy and neck patient groups will receive the training for 4 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck Pain Patients (Experimental)
  Interventions: Other: Lateralization Imagery Training
- Healty Controls (Active Comparator)
  Interventions: Other: Lateralization Imagery Training

INTERVENTIONS:
Other: Lateralization Imagery Training — Lateralization Imagery Training (LIE) is a form of implicit motor imagery that involves determining as accurately and quickly as possible whether an image of a body part belongs to the left or right side. It has been assumed that LIE performance differences reflect changes in central nervous system functioning, errors in judgment, and changes in bodily representations. It has been shown that LIE is a complex mental task that includes cognitive, sensory, motor and behavioral processes and can be associated with them. A study showed that there was a strong correlation between LIE and proprioception.
  Within the scope of our study, 3 weeks of training will be provided; Lateralization imagery training will be given every day for the first 2 weeks, and imagery training will be given 3 days a week in the 2nd and 3rd weeks. A total of 20 sessions of treatment will be applied, including 14 sessions of lateralization and 6 sessions of visualization training.

SUMMARY:
In this study, it was planned to investigate the effectiveness of lateralization and imagery training in individuals with chronic neck pain. A total of 34 individuals, 17 with chronic neck pain and 17 healthy individuals between the ages of 18-65, will be included in the study. Individuals in each group will be treated with lateralization and imagery training for 4 weeks. Before treatment, individuals' cognitive states will be evaluated with neuropsychological tests (Montreal Cognitive Assessment, Stroop test). Then, after completing the Motor Imagery Evaluation, Neck Pain Task Force Scale, Pain Severity, Kinesiophobia Evaluation, Neck Disability Evaluation, Proprioception Sense Test, Body Awareness Evaluation (Fremantle Neck Awareness Questionnaire) and Evaluation of Compliance with the Treatment Program, EEG recording of the individuals will be performed. EEG recording will be performed and analyzed with Spontaneous EEG, Oddball Paradigm and Lateralization paradigm. After four weeks of treatment, all pre-treatment tests will be repeated and then the individuals will be taken again for EEG recording. Brain oscillations will be examined through EEG analysis before and after treatment, and the extent to which brain activities have changed and the possible effect of the treatment on brain activities will be investigated.

DETAILED DESCRIPTION:
Chronic neck pain is one of the debilitating conditions that can impair the ability to perform regular daily activities, reduce productivity, and negatively impact quality of life. Approximately two-thirds of people in developed countries experience neck pain. At any given time, approximately 14% to 16% of the adult population globally experiences neck pain, with an average lifetime prevalence of 48.5%. Chronic pain is categorized as pain that lasts more than three months.

It is very important to understand neuroplasticity to know how acute pain turns into chronic pain. Local inflammation of injured tissue increases the sensitivity of peripheral sensory neurons (nociceptors), resulting in recurrent abnormal afferent input to the central nervous system. Chronic pain causes abnormal cortical reorganization and abnormal neural circuit formation in subcortical structures through neuroplastic changes in the brain. Due to chronic pain; Deterioration in body schema perception, weaknesses in perceiving somatosensory differences, deterioration in movement quality and difficulties in performing complex movements occur. Cervical afferent input to the upper centers may change for these reasons, thus cervical proprioception may be impaired.

One of the main problems of patients with neck pain is that impairment of cervical proprioception leads to impairment of cervical sensorimotor control. A study revealed that the focus of studies should be on special programs that address different aspects of sensorimotor control disorders, such as training aimed at improving proprioception and muscle coordination.

Motor imagery (MI) approach is a method created to reduce pain and improve function, especially in chronic painful situations. It is known that imagination and active movement pass through and occur through similar neural pathways. In MI, it is seen that similar regions are activated during imagination in the same way that the regions that occur during real movement and are activated in the motor cortex. In this method, premotor cortex activation is achieved without primary motor cortex activation. Movement signals are produced in cortical areas before movement is performed.

Lateralization Imagery Training (LIE) is a form of implicit motor imagery that involves determining as accurately and quickly as possible whether an image of a body part belongs to the left or right side. It has been assumed that LIE performance differences reflect changes in central nervous system functioning, errors in judgment, and changes in bodily representations. It has been shown that LIE is a complex mental task that includes cognitive, sensory, motor and behavioral processes and can be associated with them. A study showed that there was a strong correlation between LIE and proprioception.

It has been shown that individuals with chronic pain have a decrease in their ability to distinguish right-left (extremity lateralization). Being able to distinguish right from left is related to one's ability to position one's body in space. With right-left discrimination training, the higher cortical functions of the right brain hemisphere, such as whole vision, visual skills and body schema perception, are reactivated and tried to be imparted to the individual.

In some patients with chronic pain, thinking about moving the painful extremity may cause overactivation of motor-related cerebral cortices, including the cingulate motor area (SMA) and primary motor cortex, which may aggravate the cognition associated with painful experiences. For these reasons, it is an issue that needs to be investigated what kind of changes occur in patients with chronic neck pain, especially in cognitive affect and cortex activities. Electroencephalography (EEG), a non-invasive technique, is one of the methods that measure activity in the cortex. To our knowledge, there is no study in the literature investigating the effects of lateralization imagery training on EEG brain oscillations, pain intensity, kinesiophobia and proprioception in individuals with chronic neck pain.

In the light of this information, the primary purpose of the study is to a) examine whether brain activity changes at the cortex level by measuring the electrical activities in the brain during lateralization imagery training (LIE) with EEG, and b) determine whether LIE affects the severity of neck pain and disability in individuals with chronic neck pain. The aim is to examine its effects on sensory acuity, proprioception, kinesiophobia and body awareness.

The secondary aim of this study is; To evaluate the relationship between pain intensity/disability and sensory acuity, proprioception, kinesiophobia and body awareness in individuals with chronic neck pain.

The hypotheses developed to achieve these goals are; Hypothesis 1. Lateralization imagery training has an effect on brain activities in individuals with chronic neck pain.

Hypothesis 2. Lateralization imagery training has an effect on pain intensity in individuals with chronic neck pain.

Hypothesis 3. Lateralization imagery training has an effect on disability in individuals with chronic neck pain.

Hypothesis 4. Lateralization imagery training has an effect on sensory acuity (two-point discrimination) in individuals with chronic neck pain.

Hypothesis 5. Lateralization imagery training has an effect on proprioception in individuals with chronic neck pain.

Hypothesis 6. Lateralization imagery training has an effect on kinesiophobia in individuals with chronic neck pain.

Hypothesis 5. Lateralization imagery training has an effect on body awareness in individuals with chronic neck pain.

Hypothesis 7. There is a relationship between the severity of neck pain and disability and sensory acuity, proprioception, kinesiophobia and body awareness in individuals with chronic neck pain.

Material and Method: Asymptomatic individuals with chronic neck pain will be included in the study. Individuals with chronic neck pain and asymptomatic individuals will be divided into two groups: study and control, in a randomized controlled manner. Both groups will receive 3-week lateralization imagery training; Lateralization imagery training will be given every day for the first 2 weeks, and in the 2nd and 3rd weeks, imagery training will be given 3 days a week in addition to LIE. A total of 20 sessions of treatment will be applied, including 14 sessions of lateralization and 6 sessions of visualization training.

The sample size was calculated using the G*Power 3.1.9.2 analysis program. A total sample size of 34 individuals, at least 17 for both groups, was estimated with 80% power, 0.08 alpha level and 0.8 effect size.

Working Group - Neck Pain Group

Individuals with chronic neck pain can see Specialist at FSM Medical Center. Dr. Emel Deniz Şahin will be included in the working group according to the inclusion and exclusion criteria. First, initial evaluations and all tests of the included individual will be performed by the physiotherapist. Secondly, individuals will be directed to the laboratory where EEG recording will be performed. Travel expenses of individuals will be covered by the physiotherapist.

Within the scope of our study, 3 weeks of training will be provided; Lateralization imagery training will be given every day for the first 2 weeks, and imagery training will be given 3 days a week in the 2nd and 3rd weeks. A total of 20 sessions of treatment will be applied, including 14 sessions of lateralization and 6 sessions of visualization training.

It will be done in 4 stages:

Stage 1: Information about the demographic and physical characteristics of the participants will be obtained. NPT, motor imagery assessment will be performed to determine compliance with inclusion criteria. Then, pain intensity, kinesiophobia, body awareness, disability evaluation, sensory acuity, proprioception sensory tests will be applied to the individual.

Stage 2: Individuals' spontaneous EEG recording will be performed, followed by the Oddball Paradigm and then the Lateralization Imagination Paradigm recording.

Stage 3: Individuals will be given 3 weeks of training. Lateralization imagery training will be given every day for the first 2 weeks, imagery training will begin in addition to LIE in the 2nd week, and will continue in the 3rd week. Imagery training will be 6 sessions in total, 3 days a week. A total of 20 sessions of treatment will be applied, including 14 sessions of lateralization and 6 sessions of visualization training. After LIE and imagery training is completed, individuals will be evaluated for pain, kinesiophobia, neck disability index, and Montreal cognitive evaluation. Two-point discrimination sensory test, muscle activation, and proprioceptive sensory tests will be repeated.

Stage 4: After the three-week LIE and imagery training and tests are completed, spontaneous EEG recording, Oddball Paradigm, and then Lateralization Imagination Paradigm will be repeated.

Healthy Group

According to the inclusion criteria, individuals will be included in the control group. Travel expenses of individuals will be covered by the physiotherapist.

It will be done in 4 stages:

Stage 1: Information about the demographic and physical characteristics of the participants will be obtained. NPT, motor imagery assessment will be performed to determine compliance with inclusion criteria. Then, pain intensity, kinesiophobia, body awareness, disability evaluation, sensory acuity, proprioception sensory tests will be applied to the individual.

Stage 2: Individuals' spontaneous EEG recording will be performed, followed by the Oddball Paradigm and then the Lateralization Imagination Paradigm recording.

Stage 3: Individuals will be given 3 weeks of training. Lateralization imagery training will be given every day for the first 2 weeks, imagery training will begin in addition to LIE in the 2nd week and will continue in the 3rd week. Imagery training will be 6 sessions in total, 3 days a week. A total of 20 sessions of treatment will be applied, including 14 sessions of lateralization and 6 sessions of visualization training. After LIE and imagery training is completed, individuals will be evaluated for pain, kinesiophobia, neck disability index, and Montreal cognitive evaluation. Two-point discrimination sensory test, muscle activation, and proprioceptive sensory tests will be repeated.

Stage 4: After the training and tests are completed, spontaneous EEG recording, Oddball Paradigm, and then Lateralization Imagination Paradigm will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  * Between the ages of 18-65, having neck pain lasting more than 3 months,
  * Speaks and understands the Turkish language at a sufficient level,
  * Able to use telephone and computer,
  * Being literate,
  * Scored 21 or more on the Montreal Cognitive Assessment (MoCA) scale, which evaluates the cognitive status of individuals,
  * Reporting pain intensity as 30 mm or more on the Visual Analogue Scale (VAS),
  * Individuals with level 3 according to the Neck Pain Task Force Scale will be included.

Inclusion criteria for healthy group / Asymptomatic Individuals

* Asymptomatic between the ages of 18-65,
* Individuals matched with the study group in terms of body mass index and age
* Do not feel neck or back pain that prevents them from normal activities,
* Those who have not previously received medical intervention or treatment for their neck problem,
* Being literate,
* Individuals who score 21 or above on the Montreal Cognitive Assessment (MoCA) scale, which evaluates the cognitive status of individuals, will be included.

Exclusion criteria

* Have received physiotherapy treatment due to neck pain in the last 6 months,
* Those who have had neck surgery,
* Suspicion of malignant or systemic disease,
* Having a neurological disease or injury,
* Individuals with vertigo, nausea, visual disturbances will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Status Assessment (Montreal Cognitive Assessment: MoCA) | Baseline
  It will be used to evaluate the cognitive status of individuals and to exclude participants from the study. It is a test that aims to evaluate participants in 7 cognitive aspects such as attention, concentration, memory, language, calculation, spatial-visual skills, reasoning and orientation. It takes approximately ten minutes. The highest score that can be obtained from the test is 30. The cognitive level of the participant who scores 21 points or above is considered normal. Turkish validity-reliability study was conducted by Özdilek and Kenangil in 2014.
Stroop test (quick) | Baseline, and up to 4 weeks
  It is a cognitive control test consisting of three parts developed by J. R. Stroop in 1935. The Stroop task and related tests are considered the gold standard of attention measurements in the literature. In the first part of the test, subjects are presented with color names and asked to read them as quickly as possible. In the second part, you are asked to say the colors of dot clusters printed with colored ink as quickly as possible. In the third part, the students are asked to read the words written in ink of a different color than the name of the presented color as quickly (and loudly) as possible. The Turkish validity and reliability study was conducted by Karakaş et al. in 1999.
Motor Imagery Assessment | Baseline
  Made using the Movement Imagery Questionnaire-3. The Turkish validity and reliability study of the questionnaire was conducted by Dilek et al. It was made by. It consists of 3 subscales and a total of 12 items that evaluate external visual imagery, internal visual imagery, and kinesthetic imagery. Each of the 12 tasks in the survey is first performed physically, then the participant returns to the starting position and imagery is performed according to the desired type of imagery. Scoring is made between 1 and 7, with "1 point: very difficult to see/feel, 7 points: very easy to see/feel." When calculating the score, internal visual imagery, external visual imagery and kinesthetic imagery scores are added separately, divided by 4 and averaged to obtain the score of each subscale.
Pain Intensity | Baseline, and up to 4 weeks
  Individuals' pain intensity will be evaluated subjectively with the Visual Analog Scale (VAS). This scale consists of a 10 cm linear line. The starting point of the line is 0, no pain; The endpoint of 10 is the worst pain ever experienced in life; 5 indicates moderate pain. People will be asked to numerically rate the severity of their pain on the scale.
Kinesiophobia Assessment | Baseline, and up to 4 weeks
  Fear of movement will be evaluated with the TAMPA kinesiophobia scale (TKÖ). TAS is a questionnaire consisting of 17 questions developed by Korietal in 1991 for musculoskeletal pain. This scale includes parameters for injury/re-injury and fear avoidance in activities related to . In this scale, each question was scored as (1 = disagree, 4 = strongly agree). While scoring, items 4, 8, 12 and 16 are reversed and then the total score is obtained. The person receives a total score between 17-68. The Turkish reliability of the Tampa Kinesiophobia Scale was conducted by Yılmaz et al.
Evaluation of Neck Disability | Baseline, and up to 4 weeks
  The extent to which individuals' chronic neck pain affects their daily living activities will be evaluated with the Neck Disability Index (NEI). The Turkish validity and reliability of the index was determined by Telci et al. The index, which evaluates subjective symptoms and activities of daily living, consists of a total of 10 sections (pain intensity, personal care, lifting, reading, headache, concentration, work life, driving, sleep and leisure activities). There are 6 options for each section, ranging from 0 to 5 points. The total score varies between 0 and 50 (0: no disability; 50: maximum disability), and an increase in the total score indicates that the disability increases. In the evaluation in our study, the percentage of each score will be calculated to obtain an equal score distribution in case the patients do not answer some questions. 8 percent and below is considered "no excuse".
Proprioception Sense Test | Baseline, and up to 4 weeks
  Cervical joint position error will be measured using the Dualer IQ digital inclinometer (J-Tech Medical, Midvale, UT, USA). Digital inclinometer spine assessment protocols are well established and approved by the American Medical Association. Digital inclinometer allows clinicians to evaluate range of motion and proprioception using dynamic inclinometry similar to that used in other goniometric protocols. Digital inclinometer has demonstrated test-retest reliability for measuring spinal range of motion.
Body Awareness Assessment | Baseline, and up to 4 weeks
  Individuals' neck awareness will be assessed with the Fremantle Neck Awareness Questionnaire. Developed by Benedict Wand, its Turkish validity and reliability were confirmed by Onan et al. Likert type assessing individual-specific altered perception (0 = I never/never feel like this, 1= I rarely feel like this, 2 = Sometimes, or some of the time I feel like this, 3 = I often feel like this, 4 = I always or most of the time feel like this) It is a simple survey. The survey asks individuals 9 questions, such as how they perceive their neck in relation to their body and how they perceive their body position.
EEG power in alpha, theta, beta band | Baseline, and up to 4 weeks
  Evaluation of brain oscillations with EEG analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ülger, Prof, Study Director — Hacettepe University; Bahar Güntekin, Prof, Study Director — Medipol University; Ayşenur Zaim, Master (Canditate), Principal Investigator — Medipol University; Ayşegül Bostan, PhD (Candidate), Principal Investigator — Hacettepe University
Locations (1):
- Bahcesehir Universty, Istanbul, BESIKTAS, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carvalho, R.Cd., Maglioni, C.B., Machado, G.B., Araújo, J.Ed., Silva, J.R.Td., Silva, M.Ld. 2018.
- [Background] Genebra CVDS, Maciel NM, Bento TPF, Simeao SFAP, Vitta A. Prevalence and factors associated with neck pain: a population-based study. Braz J Phys Ther. 2017 Jul-Aug;21(4):274-280. doi: 10.1016/j.bjpt.2017.05.005. Epub 2017 May 20. PMID 28602744
- [Background] Hague M, Shenker N. How to investigate: Chronic pain. Best Pract Res Clin Rheumatol. 2014 Dec;28(6):860-74. doi: 10.1016/j.berh.2015.04.005. Epub 2015 May 23. PMID 26096090
- [Background] Brumagne S, Diers M, Danneels L, Moseley GL, Hodges PW. Neuroplasticity of Sensorimotor Control in Low Back Pain. J Orthop Sports Phys Ther. 2019 Jun;49(6):402-414. doi: 10.2519/jospt.2019.8489. PMID 31151373
- [Background] Yam MF, Loh YC, Tan CS, Khadijah Adam S, Abdul Manan N, Basir R. General Pathways of Pain Sensation and the Major Neurotransmitters Involved in Pain Regulation. Int J Mol Sci. 2018 Jul 24;19(8):2164. doi: 10.3390/ijms19082164. PMID 30042373
- [Background] Schwoebel J, Coslett HB, Bradt J, Friedman R, Dileo C. Pain and the body schema: effects of pain severity on mental representations of movement. Neurology. 2002 Sep 10;59(5):775-7. doi: 10.1212/wnl.59.5.775. PMID 12221179
- [Background] Reddy RS, Tedla JS, Dixit S, Abohashrh M. Cervical proprioception and its relationship with neck pain intensity in subjects with cervical spondylosis. BMC Musculoskelet Disord. 2019 Oct 15;20(1):447. doi: 10.1186/s12891-019-2846-z. PMID 31615495
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control. Man Ther. 2008 Feb;13(1):2-11. doi: 10.1016/j.math.2007.06.003. Epub 2007 Aug 16. PMID 17702636
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control--Part 2: case studies. Man Ther. 2008 Jun;13(3):266-75. doi: 10.1016/j.math.2007.11.002. Epub 2008 Jan 3. PMID 18180194
- [Background] Peng B, Yang L, Li Y, Liu T, Liu Y. Cervical Proprioception Impairment in Neck Pain-Pathophysiology, Clinical Evaluation, and Management: A Narrative Review. Pain Ther. 2021 Jun;10(1):143-164. doi: 10.1007/s40122-020-00230-z. Epub 2021 Jan 12. PMID 33464539
- [Background] Jeannerod, M. 1994. "The representing brain: Neural correlates of motor intention and imagery", Cambridge University Press, 187-202.
- [Background] Hetu S, Gregoire M, Saimpont A, Coll MP, Eugene F, Michon PE, Jackson PL. The neural network of motor imagery: an ALE meta-analysis. Neurosci Biobehav Rev. 2013 Jun;37(5):930-49. doi: 10.1016/j.neubiorev.2013.03.017. Epub 2013 Apr 10. PMID 23583615
- [Background] Solodkin A, Hlustik P, Chen EE, Small SL. Fine modulation in network activation during motor execution and motor imagery. Cereb Cortex. 2004 Nov;14(11):1246-55. doi: 10.1093/cercor/bhh086. Epub 2004 May 27. PMID 15166100
- [Background] Osuagwu BA, Vuckovic A. Similarities between explicit and implicit motor imagery in mental rotation of hands: an EEG study. Neuropsychologia. 2014 Dec;65:197-210. doi: 10.1016/j.neuropsychologia.2014.10.029. Epub 2014 Oct 30. PMID 25446966
- [Background] Moseley, G.L. 2012. "The Graded Motor Imagery Handbook", Noigroup publications, Australia.
- [Background] Pelletier R, Bourbonnais D, Higgins J, Mireault M, Danino MA, Harris PG. Left Right Judgement Task and Sensory, Motor, and Cognitive Assessment in Participants with Wrist/Hand Pain. Rehabil Res Pract. 2018 Aug 26;2018:1530245. doi: 10.1155/2018/1530245. eCollection 2018. PMID 30225144
- [Background] Elsig S, Luomajoki H, Sattelmayer M, Taeymans J, Tal-Akabi A, Hilfiker R. Sensorimotor tests, such as movement control and laterality judgment accuracy, in persons with recurrent neck pain and controls. A case-control study. Man Ther. 2014 Dec;19(6):555-61. doi: 10.1016/j.math.2014.05.014. Epub 2014 Jun 10. PMID 24957711
- [Background] Breckenridge, J., Ginn, K., Wallwork, S., McAuley, J. 2016. " Does Upper Limb Pain Affect the Left/Right Judgment Task? A Systematic Review and Meta-analysis", HAND, 2016(11), 136.
- [Background] Adın, R.M., Kuru Ç.A. 2018. "Aşamalı Motor İmgeleme Yaklaşımı/Graded Motor Imagery Approach", In book: Fizyoterapi Seminerleri E Kitap, 17-23.
- [Background] Osumi M, Sumitani M, Nishi Y, Nobusako S, Dilek B, Morioka S. Fear of movement-related pain disturbs cortical preparatory activity after becoming aware of motor intention. Behav Brain Res. 2021 Aug 6;411:113379. doi: 10.1016/j.bbr.2021.113379. Epub 2021 May 26. PMID 34051229
- [Background] Wolpaw JR, Loeb GE, Allison BZ, Donchin E, do Nascimento OF, Heetderks WJ, Nijboer F, Shain WG, Turner JN. BCI Meeting 2005--workshop on signals and recording methods. IEEE Trans Neural Syst Rehabil Eng. 2006 Jun;14(2):138-41. doi: 10.1109/TNSRE.2006.875583. PMID 16792279
- [Background] Ozdilek B, Kenangil G. Validation of the Turkish Version of the Montreal Cognitive Assessment Scale (MoCA-TR) in patients with Parkinson's disease. Clin Neuropsychol. 2014;28(2):333-43. doi: 10.1080/13854046.2014.881554. Epub 2014 Feb 17. PMID 24528299
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Manna, C.G., et al. 2011. Sayfa 392-304. "Benton Visual Retention Test in Encyclopedia of Clinical Neuropsychology", Editors: Kreutzer, J.S., DeLuca, J., Caplan, B. New York: Springer.
- [Background] Stroop, J.R. 1935. "Studies of interference in serial verbal reactions", Journal of experimental psychology, 18, 643.
- [Background] MacLeod, C.M. 1992. "The Stroop task: The
- [Background] Karakaş, S., Irak, M., Ersezgin, Ö. 1998. "Wisconsin Kart Eşleme Testi (WCST) ve Stroop Testi TBAG formu puanlarının test içi ve testler-arası ilişkileri", X Ulusal Psikoloji Kongresi özet kitabı, 44.
- [Background] Dilek, B., Ayhan, C., Yakut, Y. 2020. "Reliability and validity of the Turkish version of the movement imagery questionnaire-3: Its cultural adaptation and psychometric properties", Neurol Sci Neurophysiol, 37, 221-227.
- [Background] Haldeman S, Carroll L, Cassidy JD, Schubert J, Nygren A; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. The Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders: executive summary. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S5-7. doi: 10.1097/BRS.0b013e3181643f40. No abstract available. PMID 18204400
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] Yılmaz, Ö.T., Yakut, Y., Uygur, F., Uluğ, N. 2011. "Tampa kinezyofobi ölçeği"nin Türkçe versiyonu ve test-tekrar test güvenirliği", Fizyoterapi Rehabilitasyon, 22(1), 44-49.
- [Background] Telci EA, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagli N. The cultural adaptation, reliability, and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2009 Jul 15;34(16):1732-5. doi: 10.1097/BRS.0b013e3181ac9055. PMID 19770615
- [Background] Harvie DS, Kelly J, Buckman H, Chan J, Sutherland G, Catley M, Novak J, Tuttle N, Sterling M. Tactile acuity testing at the neck: A comparison of methods. Musculoskelet Sci Pract. 2017 Dec;32:23-30. doi: 10.1016/j.msksp.2017.07.007. Epub 2017 Jul 29. PMID 28800436
- [Background] Öksüz, Ç., Akel, B.S. 2016. Sayfa 299-312. Fizyoterapi ve Rehabilitasyon Cilt 1. Editör: Karaduman A.A., Yılmaz Ö.T. Ankara: Hipokrat Kitabevi ve Pelikan Kitabevi.
- [Background] Nitschke JE, Nattrass CL, Disler PB, Chou MJ, Ooi KT. Reliability of the American Medical Association guides' model for measuring spinal range of motion. Its implication for whole-person impairment rating. Spine (Phila Pa 1976). 1999 Feb 1;24(3):262-8. doi: 10.1097/00007632-199902010-00013. PMID 10025021
- [Background] Tousignant M, Boucher N, Bourbonnais J, Gravelle T, Quesnel M, Brosseau L. Intratester and intertester reliability of the Cybex electronic digital inclinometer (EDI-320) for measurement of active neck flexion and extension in healthy subjects. Man Ther. 2001 Nov;6(4):235-41. doi: 10.1054/math.2001.0419. PMID 11673934
- [Background] Santos, C.M.D., Ferreira, G., Malacco, P.L., Sabino, G.S., Moraes, G.F.D.S., Felício, D.C. 2012. "Intra and inter examiner reliability and measurement error of goniometer and digital inclinometer use", Revista Brasileira de Medicina do Esporte, 18, 38-41.
- [Background] Wand BM, Catley MJ, Rabey MI, O'Sullivan PB, O'Connell NE, Smith AJ. Disrupted Self-Perception in People With Chronic Low Back Pain. Further Evaluation of the Fremantle Back Awareness Questionnaire. J Pain. 2016 Sep;17(9):1001-12. doi: 10.1016/j.jpain.2016.06.003. Epub 2016 Jun 18. PMID 27327235
- [Background] Onan D, Gokmen D, Ulger O. The Fremantle Neck Awareness Questionnaire in Chronic Neck Pain Patients: Turkish Version, Validity and Reliability Study. Spine (Phila Pa 1976). 2020 Feb 1;45(3):E163-E169. doi: 10.1097/BRS.0000000000003207. PMID 31425430
- [Background] Cadmus-Bertram L, Irwin M, Alfano C, Campbell K, Duggan C, Foster-Schubert K, Wang CY, McTiernan A. Predicting adherence of adults to a 12-month exercise intervention. J Phys Act Health. 2014 Sep;11(7):1304-12. doi: 10.1123/jpah.2012-0258. Epub 2013 Oct 31. PMID 24176780
- [Background] Moseley GL. Graded motor imagery for pathologic pain: a randomized controlled trial. Neurology. 2006 Dec 26;67(12):2129-34. doi: 10.1212/01.wnl.0000249112.56935.32. Epub 2006 Nov 2. PMID 17082465
- [Background] Priganc VW, Stralka SW. Graded motor imagery. J Hand Ther. 2011 Apr-Jun;24(2):164-8; quiz 169. doi: 10.1016/j.jht.2010.11.002. Epub 2011 Feb 9. PMID 21306870
- [Background] Moseley GL. Why do people with complex regional pain syndrome take longer to recognize their affected hand? Neurology. 2004 Jun 22;62(12):2182-6. doi: 10.1212/01.wnl.0000130156.05828.43. PMID 15210879
- [Background] Wallwork SB, Butler DS, Fulton I, Stewart H, Darmawan I, Moseley GL. Left/right neck rotation judgments are affected by age, gender, handedness and image rotation. Man Ther. 2013 Jun;18(3):225-30. doi: 10.1016/j.math.2012.10.006. Epub 2013 Jan 26. PMID 23357411
- [Background] Sur S, Sinha VK. Event-related potential: An overview. Ind Psychiatry J. 2009 Jan;18(1):70-3. doi: 10.4103/0972-6748.57865. PMID 21234168
- [Background] Amin HU, Malik AS, Kamel N, Chooi WT, Hussain M. P300 correlates with learning & memory abilities and fluid intelligence. J Neuroeng Rehabil. 2015 Sep 23;12:87. doi: 10.1186/s12984-015-0077-6. PMID 26400233
- [Background] Huettel SA, McCarthy G. What is odd in the oddball task? Prefrontal cortex is activated by dynamic changes in response strategy. Neuropsychologia. 2004;42(3):379-86. doi: 10.1016/j.neuropsychologia.2003.07.009. PMID 14670576
- [Background] Stevens AA, Skudlarski P, Gatenby JC, Gore JC. Event-related fMRI of auditory and visual oddball tasks. Magn Reson Imaging. 2000 Jun;18(5):495-502. doi: 10.1016/s0730-725x(00)00128-4. PMID 10913710
- [Background] Fukami, T., Shimada, T., Akatsuka, T., Ishikawa, F., Ishikawa B., Saito Y. 2003.
- [Background] Fajkus J, Mikl M, Shaw DJ, Brazdil M. An fMRI investigation into the effect of preceding stimuli during visual oddball tasks. J Neurosci Methods. 2015 Aug 15;251:56-61. doi: 10.1016/j.jneumeth.2015.05.005. Epub 2015 May 16. PMID 25989317